CLINICAL TRIAL: NCT02318251
Title: Stress Urinary Incontinence Physiotherapy (SUIP) - A Randomized Controlled Trial With 6-Months Follow-up
Brief Title: Stress Urinary Incontinence Physiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bern University of Applied Sciences (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Lorenz Radlinger, Prof. Dr. Lorenz Radlinger, Bern University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SUIP
Record Dates: First submitted 2014-12-04; First posted 2014-12-17 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Urinary Incontinence, Stress
Keywords: Power, rate of force development; involuntary; reflexive
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Involuntary muscle contractions (Experimental): Standard physiotherapy program (focus on involuntary reflexive pelvic floor muscle contractions)
  Interventions: Other: Involuntary muscle contractions
- Voluntary muscle contractions (Active Comparator): Physiotherapy program (focus on voluntary pelvic floor muscle contractions)
  Interventions: Other: Voluntary muscle contractions

INTERVENTIONS:
Other: Involuntary muscle contractions — Physiotherapy program focusing on involuntary pelvic floor muscle fast contractions: 9 individual physiotherapies taking place within 16 weeks. During these 16 weeks the participants will perform a home program 3x/week (3x/day) during week 1-5 and 3x/week (1x/day) in week 6-16. In the following 6 months they will perform the home program 3x/week (1x/day). This program includes the standard physiotherapy.
  Arms: Involuntary muscle contractions
Other: Voluntary muscle contractions — Physiotherapy program (physiotherapy standard program) focusing on voluntary fast contractions: 9 individual physiotherapies taking place within 16 weeks. During these 16 weeks the participants will perform a home program 3x/week (3x/day) during week 1-5 and 3x/week (1x/day) in week 6-16. In the following 6 months they will perform the home program 3x/week (1x/day).
  Arms: Voluntary muscle contractions

SUMMARY:
The purpose of the present study is to compare two different physiotherapy programs regarding their effect on stress urinary incontinence.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI), the most prevalent type of urinary incontinence, is defined as involuntary loss of urine during effort, or physical exertion (e.g. sporting activities), or upon sneezing, or coughing (Haylen et al, 2010). The overall prevalence of stress, urge, mixed, and any UI was 23.7%, 9.9%, 14.5%, and 49.2%, respectively (Minassian et al, 2008).

Numerous epidemiologic studies show that parity is a risk factor for SUI. Other significant risk factors are age, weight, obesity, chronic pulmonary diseases, ethnic background, and menopause. (Minassian et al, 2008; Matthews et al, 2013) Urinary incontinence affects four times more women (51.1%) than men (13.9%) (Markland et al, 2011). It has an impact on the physical, psychosocial, social, personal, and economic well-being of the affected individuals and of their families. It is associated with a concomitant impairment of activities and participation, and a higher risk of suffering from anxiety disorders has been shown. (Goldstick & Constantini, 2014; Hunskaar et al, 2003).

SUI is increasingly recognized as a health and economic problem, which not only troubles the affected women, but also implies a substantial economic burden on the health and social services (Hampel et al, 2004).

Consequently, as physiotherapy has proven to be good value for the money, its effectiveness could contribute to a reduction in the cost of health care.

Pelvic floor muscles (PFM) have to be able to contract strongly (Shishido et al, 2008), rapidly and reflexively (Deffieux et al; 2008; Morin et al, 2004) to guarantee continence. The ability of PFM to generate rapid and strong contractions results in the generation of an adequate squeeze pressure in the proximal urethra, which maintains a pressure higher than that in the bladder, thus preventing leakage (Miller et al, 1994). Rapid and reflexive PFM contractions are crucial for maintaining continence, preceding an abrupt rise in the intra-abdominal pressure associated with coughing, sneezing, running, or jumping (Morin et al., 2004). Studies have shown that the PFM function regarding power (rate of force development) was impaired in incontinent women compared to continent women (Deffieux et al, 2008; Morin et al, 2004).

PFM training - defined as a program of repeated voluntary PFM contractions taught and supervised by a health care professional - is the most commonly used physiotherapy treatment for women with SUI and is effective in the treatment of female stress and mixed urinary incontinence and, therefore, is recommended as a first-line therapy (Dumoulin et al, 2014; Bø, 2012). As recommended by the International Consultation on Incontinence (ICI) PFM training should generally be the first step of treatment before surgery (Abrams et al, 2010). However, standard SUI physiotherapy concentrates on voluntary contractions even though the situations provoking SUI such as sneezing, coughing, jumping and running (Haylen et al, 2010) require involuntary fast reflexive pelvic floor muscle contractions. Although training procedures following the concepts of training science and sports medicine are generally well known and widely implemented in rehabilitation and sports (ACSM, 2009; Schmidtbleicher & Gollhofer, 1991), the optimal, and well standardized training protocol for involuntary, fast, and reflexive PFM contractions still remains unknown.

Consequently, the research group developed a standardized therapy program, which includes the standard therapy and additionally focuses on involuntary fast reflexive PFM contractions. The additional exercises are well known and applied in physiotherapy, however not yet regarding SUI.

Therefore, the aim of the present study is to compare two different physiotherapy programs for women suffering from SUI. Both programs include standard physiotherapy. Both follow the concepts of training science (periodization/ exercise sequence and training of specific muscle strength components). One program focuses on voluntary fast contractions (standard physiotherapy; control group), the other one focuses on involuntary fast reflexive PFM contractions (experimental group).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Stress urinary incontinence (based on the patient's history)
* Mixed incontinence (with dominant SUI)
* 1 year post-partal, parous, nulliparous, pre- or post-menopausal
* BMI 18-30
* Participants must be medically and physically fit for the exercises (running, jumps)
* Stable on systemic or local estrogen treatment for the past 3 months prior to inclusion

Exclusion Criteria:

* Urge incontinence or predominant urgency in incontinence
* Prolapse > grade 1 POP-Q (Bump et al., 1996) (uterus, cystocele, rectocele during Valsalva maneuver)
* Pregnancy (test to accomplish)
* Current urinary tract or vaginal infection
* Menstruation on the day of examination
* Lactation period not yet finished
* Contraindications for measurements, e.g. acute inflammatory or infectious disease, tumor, fracture
* De novo systemic or local estrogen treatment (< 3 months)
* De novo drug treatment with anticholinergics or other bladder active substances (tricyclic antidepressants, Selective Serotonin Reuptake Inhibitor etc.)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-01; Primary Completion 2018-06-30 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
International Consultation on Incontinence Modular Questionnaire - Urinary Incontinence short form (ICIQ-UIsf (short form)) | up to 6 months follow up
  The ICIQ-UIsf provides a brief and robust measure to assess the impact of symptoms of incontinence on quality of life and outcome of treatment

SECONDARY OUTCOMES:
Pelvic floor muscle electromyography | up to 6 months follow up
  Electromyography (EMG) activity measurements during rest, during maximal Voluntary contraction, fast voluntary contractions and during involuntary contractions (squat jumps, counter movement jumps, drop jumps), and during running at 7,9,11 km/h)
20-minute PAD-test | up to 6 months follow up
  The 20 min Pad Test assesses urine loss and leakage volume of the participant
International Consultation on Incontinence Modular Questionnaire - Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTSqol) | up to 6 months follow up
  The ICIQ-LUTSqol questionnaire evaluates the impact the participant's quality of life, with reference also to social effects
International Consultation on Incontinence Modular Questionnaire - Urinary Incontinence short form (ICIQ-UIsf (short form)) | At the 6 months follow up
  See primary outcome

OTHER OUTCOMES:
Pelvic floor manual muscle testing | up to 6 months follow up
  Pelvic floor muscle strength will be digitally assessed by the Oxford grading scale.
Home exercise adherence | up to 6 months follow up
  Adherence to the home exercise program will be assessed, i.e. how many of the total of therapy sessions will be completed individually

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Radlinger, Prof. Dr., Study Director — Bern University of Applied Sciences; Kuhn Annette, PD Dr. med., Study Director — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Hospital, Inselspital, Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Minassian VA, Stewart WF, Wood GC. Urinary incontinence in women: variation in prevalence estimates and risk factors. Obstet Gynecol. 2008 Feb;111(2 Pt 1):324-31. doi: 10.1097/01.AOG.0000267220.48987.17. PMID 18238969
- [Background] Matthews CA, Whitehead WE, Townsend MK, Grodstein F. Risk factors for urinary, fecal, or dual incontinence in the Nurses' Health Study. Obstet Gynecol. 2013 Sep;122(3):539-45. doi: 10.1097/AOG.0b013e31829efbff. PMID 23921863
- [Background] Markland AD, Richter HE, Fwu CW, Eggers P, Kusek JW. Prevalence and trends of urinary incontinence in adults in the United States, 2001 to 2008. J Urol. 2011 Aug;186(2):589-93. doi: 10.1016/j.juro.2011.03.114. PMID 21684555
- [Background] Goldstick O, Constantini N. Urinary incontinence in physically active women and female athletes. Br J Sports Med. 2014 Feb;48(4):296-8. doi: 10.1136/bjsports-2012-091880. Epub 2013 May 18. PMID 23687004
- [Background] Hunskaar S, Burgio K, Diokno A, Herzog AR, Hjalmas K, Lapitan MC. Epidemiology and natural history of urinary incontinence in women. Urology. 2003 Oct;62(4 Suppl 1):16-23. doi: 10.1016/s0090-4295(03)00755-6. PMID 14550833
- [Background] Hampel C, Artibani W, Espuna Pons M, Haab F, Jackson S, Romero J, Gavart S, Papanicolaou S. Understanding the burden of stress urinary incontinence in Europe: a qualitative review of the literature. Eur Urol. 2004 Jul;46(1):15-27. doi: 10.1016/j.eururo.2004.02.003. PMID 15183544
- [Background] Shishido K, Peng Q, Jones R, Omata S, Constantinou CE. Influence of pelvic floor muscle contraction on the profile of vaginal closure pressure in continent and stress urinary incontinent women. J Urol. 2008 May;179(5):1917-22. doi: 10.1016/j.juro.2008.01.020. Epub 2008 Mar 18. PMID 18353401
- [Background] Deffieux X, Hubeaux K, Porcher R, Ismael SS, Raibaut P, Amarenco G. Abnormal pelvic response to cough in women with stress urinary incontinence. Neurourol Urodyn. 2008;27(4):291-6. doi: 10.1002/nau.20506. PMID 17803192
- [Background] Morin M, Bourbonnais D, Gravel D, Dumoulin C, Lemieux MC. Pelvic floor muscle function in continent and stress urinary incontinent women using dynamometric measurements. Neurourol Urodyn. 2004;23(7):668-74. doi: 10.1002/nau.20069. PMID 15382183
- [Background] Miller J, Kasper C, Sampselle C. Review of muscle physiology with application to pelvic muscle exercise. Urol Nurs. 1994 Sep;14(3):92-7. No abstract available. PMID 7732424
- [Background] Dumoulin C, Hay-Smith EJ, Mac Habee-Seguin G. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2014 May 14;(5):CD005654. doi: 10.1002/14651858.CD005654.pub3. PMID 24823491
- [Background] Bo K. Pelvic floor muscle training in treatment of female stress urinary incontinence, pelvic organ prolapse and sexual dysfunction. World J Urol. 2012 Aug;30(4):437-43. doi: 10.1007/s00345-011-0779-8. Epub 2011 Oct 9. PMID 21984473
- [Background] Abrams P, Avery K, Gardener N, Donovan J; ICIQ Advisory Board. The International Consultation on Incontinence Modular Questionnaire: www.iciq.net. J Urol. 2006 Mar;175(3 Pt 1):1063-6; discussion 1066. doi: 10.1016/S0022-5347(05)00348-4. PMID 16469618
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Background] Schmidtbleicher D, Gollhofer A. [Specific methods of strength training also in rehabilitation]. Sportverletz Sportschaden. 1991 Sep;5(3):135-41. doi: 10.1055/s-2007-993577. German. PMID 1759194
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322
- [Derived] Luginbuehl H, Lehmann C, Baeyens JP, Kuhn A, Radlinger L. Involuntary reflexive pelvic floor muscle training in addition to standard training versus standard training alone for women with stress urinary incontinence: study protocol for a randomized controlled trial. Trials. 2015 Nov 17;16:524. doi: 10.1186/s13063-015-1051-0. PMID 26573847